CLINICAL TRIAL: NCT07090603
Title: Age-Related Differences in Skeletal Muscle Endurance Responses to Various Relative Loads of Dynamic Resistance Exercise With and Without Peripheral Blood Flow Occlusion
Brief Title: The Effects of Age on Muscle Endurance During Resistance Exercise With and Without Blood Flow Restriction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Cameron Mitchell, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H25-01532
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Ageing; Muscle Fatigue Caused by Repetitive Muscle Exercise
Keywords: muscle endurance; muscle contraction; critical occluding tension; muscle oxygenation; NIRS; ageing; muscle fatigue; contraction induced occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Young cohort (Experimental): Young, healthy participants aged 19-35 will perform maximum repetitions of knee extension exercise at 20%, 30%, 40%, 50%, 60% and 70% of their one rep max with and without blood flow occlusion.
  Interventions: Other: Knee extension exercise
- Older cohort (Experimental): Older, healthy participants aged 65 years and up will perform maximum repetitions of knee extension exercise at 20%, 30%, 40%, 50%, 60% and 70% of their one rep max with and without blood flow occlusion.
  Interventions: Other: Knee extension exercise

INTERVENTIONS:
Other: Knee extension exercise — Maximum repetitions of knee extension exercise at 20%, 30%, 40%, 50%, 60% and 70% of participants one rep max with and without blood flow occlusion

SUMMARY:
The purpose of this study is to learn how aging affects muscle endurance during resistance exercise, and how oxygen delivery to the muscles plays a role in these changes. To answer this question, we are comparing how many repetitions of a leg exercise (knee extensions) younger and older adults can do at different exercise intensities. We will also look at how the muscles use oxygen during these exercises.

Participants will take part in 12 different exercise sessions. In each session, they will perform as many knee extensions as possible using different amounts of weight-consisting of 20%, 30%, 40%, 50%, 60% and 70% of the maximum weight they can lift one time. Each weight will be tested both with and without a cuff on the leg that temporarily reduces blood flow to the muscle.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and communicate in English
* 19-35 years of age
* 65 years of age or older
* All "No" answers on the CSEP Get Active questionnaire or doctors' approval to participate

Exclusion Criteria:

* BMI lower than 18 or greater than 32
* Current use of cigarettes or other nicotine devices
* Any major uncontrolled cardiovascular, muscular, metabolic, and/or neurological disorders
* Any medical condition impacting the ability to participate in maximal exercise
* Type one or type two diabetes
* Diagnosis of cancer or undergoing cancer treatment in the past 12 months
* Taking blood-thinning medication or the presence of a bleeding disorder
* Drug therapy with any drugs that alter skeletal muscle metabolism (i.e., Metformin, Benzodiazepines)
* Lowest calculated exercise testing load is less than the lightest weight able to be provided by the lab gymnasium equipment
* In the past six months, completing more than 300 minutes of moderate physical activity or 150 minutes of vigorous physical activity per week
* In the past six months, completing less than 150 minutes of moderate physical activity or 75 minutes of vigorous physical activity

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Maximum repetitions performed during knee extension exercise | From enrollment to the end of the final study visit (~4 weeks)
  The primary outcome of the study will be the maximum number of knee extension repetitions that participants are able to perform at varying resistive exercise loads.

SECONDARY OUTCOMES:
Local muscle tissue oxygenation during knee extension exercise | From enrollment to the end of the final study visit (~ 4 weeks)
  Muscle tissue oxygenation status will be assessed during each knee extension exercise intervention using oxygen sensors placed on the outside of the thigh.

CONTACTS AND LOCATIONS:
Overall Officials: Cameron J Mitchell, PhD (Kinesiology), Principal Investigator — University of British Columbia
Locations (1):
- Chan Gunn Pavilion, Vancouver, British Columbia, Canada